CLINICAL TRIAL: NCT03224884
Title: A Randomized Comparison Between Interscalene and Supraclavicular Brachial Plexus Blocks For Arthroscopic Shoulder Surgery
Brief Title: Interscalene Block Versus Supraclavicular Block for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Clinical Instructor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 888/17
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Pain, Postoperative; Shoulder Pain; Surgical Procedure, Unspecified; Diaphragmatic Paralysis
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Respiratory Paralysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block (Active Comparator): Patients randomized to receive an interscalene block .
  Interventions: Procedure: Interscalene block
- Supraclavicular block (Experimental): Patients randomized to receive a supraclavicular block.
  Interventions: Procedure: Supraclavicular block

INTERVENTIONS:
Procedure: Interscalene block — Ultrasound guided brachial plexus block injecting 20 mL of 0.5% levobupivacaine with 5 micrograms of epinephrine per mL in the interscalene groove, under the prevertebral fascia.
  Arms: Interscalene block
Procedure: Supraclavicular block — Ultrasound guided brachial plexus injecting 20 mL of 0.5% levobupivacaine with 5 micrograms of epinephrine per mL (3 mL in the "corner pocket" followed by 17 mL posterolateral to the brachial plexus).
  Arms: Supraclavicular block

SUMMARY:
Interscalene brachial plexus block constitutes the analgesic criterion standard for shoulder surgery. However it is associated with a high incidence of hemidiaphragmatic paralysis (HDP) that may not be tolerated by patients with chronic pulmonary disease.

This randomized controlled trial will compare ultrasound-guided interscalene block (ISB) and supraclavicular block in patients undergoing arthroscopic shoulder surgery.

The main outcome is static pain at 30 minutes after arrival in the post anesthesia care unit (PACU) as measured by a numerical rate scale (NRS) from 0 to 10.

Our research hypothesis is that interscalene and supraclavicular blocks will result in equivalent postoperative analgesia at 30 minutes in the PACU. The equivalence margin is set at 2 points

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic shoulder surgery
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy
* Coagulopathy
* Obstructive or restrictive pulmonary disease
* Renal failure
* Hepatic failure
* Allergy to local anesthetics
* Pregnancy
* Prior surgery in the corresponding side of the neck or supraclavicular fossa
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Static pain at 30 minutes after arrival in the PACU | 30 minutes
  Evaluated with a NRS from 0 to 10.

SECONDARY OUTCOMES:
Static pain at 60 minutes after arrival in the PACU | 60 minutes
  Evaluated with a NRS from 0 to 10.
Postoperative static pain at 2 hours | 2 hours
  Evaluated with a NRS from 0 to 10.
Postoperative static pain at 3 hours | 3 hours
  Evaluated with a NRS from 0 to 10.
Postoperative static pain at 6 hours | 6 hours
  Evaluated with a NRS from 0 to 10.
Postoperative static pain at 12 hours | 12 hours
  Evaluated with a NRS from 0 to 10.
Postoperative static pain at 24 hours | 24 hours
  Evaluated with a NRS from 0 to 10.
Incidence of HDP at 30 minutes after interscalene or supraclavicular block | 30 minutes post injection
  Ultrasound diagnosed HDP
Incidence of HDP at 30 minutes after arrival to PACU. | 30 minutes after arrival to PACU
  Ultrasound diagnosed HDP
Block performance time | 1 hour before surgery
  Time from skin desinfection until the end of local anesthetic injection.
Sensory and Motor block | 30 minutes post injection
  Sensorimotor block assessed every 5 minutes until 30 minutes using a 8-point composite score.
Incidence of complete block | 30 minutes post injection
  Percentage of blocks with a minimal sensorimotor composite score of 6 points out of a maximum of 8 points at 30 minutes post injection.
Procedural pain during blocks | 1 hour before surgery
  Evaluated with a NRS from 0 to 10.
Onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 6 points out of a maximum of 8 points.
Intraoperative opioid requirements | Intraoperative period
  Total amount of fentanyl required during general anesthesia.
Surgical duration | intraoperative period
  Time between skin incision and closure.
Postoperative opioid consumption | 24 hours after surgery
  Total amount of morphine required during the first 24 hours after surgery.
Patient satisfaction | 24 hours after surgery
  Patient satisfaction measured using a NRS 0 to 10 (0 = unsatisfied; 10 = very satisfied).
Block- and opioid-related side effects | 1 week
  Incidence of side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Result] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Result] Ryu T, Kil BT, Kim JH. Comparison Between Ultrasound-Guided Supraclavicular and Interscalene Brachial Plexus Blocks in Patients Undergoing Arthroscopic Shoulder Surgery: A Prospective, Randomized, Parallel Study. Medicine (Baltimore). 2015 Oct;94(40):e1726. doi: 10.1097/MD.0000000000001726. PMID 26448030
- [Result] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Result] Renes SH, Spoormans HH, Gielen MJ, Rettig HC, van Geffen GJ. Hemidiaphragmatic paresis can be avoided in ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):595-9. doi: 10.1097/aap.0b013e3181bfbd83. PMID 19916254
- [Result] Tran DQ, Dugani S, Finlayson RJ. A randomized comparison between ultrasound-guided and landmark-based superficial cervical plexus block. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):539-43. doi: 10.1097/AAP.0b013e3181faa11c. PMID 20975470
- [Result] Spence BC, Beach ML, Gallagher JD, Sites BD. Ultrasound-guided interscalene blocks: understanding where to inject the local anaesthetic. Anaesthesia. 2011 Jun;66(6):509-14. doi: 10.1111/j.1365-2044.2011.06712.x. PMID 21568985
- [Result] Lloyd T, Tang YM, Benson MD, King S. Diaphragmatic paralysis: the use of M mode ultrasound for diagnosis in adults. Spinal Cord. 2006 Aug;44(8):505-8. doi: 10.1038/sj.sc.3101889. Epub 2005 Dec 6. PMID 16331304
- [Derived] Aliste J, Bravo D, Fernandez D, Layera S, Finlayson RJ, Tran DQ. A Randomized Comparison Between Interscalene and Small-Volume Supraclavicular Blocks for Arthroscopic Shoulder Surgery. Reg Anesth Pain Med. 2018 Aug;43(6):590-595. doi: 10.1097/AAP.0000000000000767. PMID 29630033